CLINICAL TRIAL: NCT02930044
Title: Prospective Comparison of Early Subcutaneous Insulin Glargine Plus Standard of Care Versus Standard of Care for Treatment of Diabetic Ketoacidosis in the Emergency Department
Brief Title: Early Subcutaneous Insulin Glargine Plus Standard of Care for Treatment of Diabetic Ketoacidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, George Willis, MD FACEP, Director of Undergraduate Medical Education, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00070969
Record Dates: First submitted 2016-09-14; First posted 2016-10-11 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Ketoacidosis
Keywords: Emergency department; Insulin; Adult
MeSH Terms: conditions — Diabetic Ketoacidosis; Emergencies; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early glargine dose (Experimental): Subcutaneous insulin glargine will be administered within two hours of starting the IV insulin infusion.
  Interventions: Other: Early administration of subcutaneous insulin glargine dose; Other: IV insulin infusion; Drug: IV fluid repletion
- Standard therapy (Placebo Comparator): Retrospective arm that received standard insulin therapy for treatment of DKA
  Interventions: Other: IV insulin infusion; Drug: IV fluid repletion

INTERVENTIONS:
Other: Early administration of subcutaneous insulin glargine dose — DKA patients in the prospective intervention arm will receive subcutaneous glargine within two hours of starting their intravenous insulin infusion. The dose of glargine is 0.3 units/kg with a maximum dose of 30 units.
  Arms: Early glargine dose
Other: IV insulin infusion — All patients will receive the standard of care which is a protocol based continuous insulin infusion
Drug: IV fluid repletion — 0.9% NaCl or Plasmalyte A will be initiated as a continuous infusion for volume repletion. Fluids will be switched to contain potassium if serum potassium is less than 3.3 mEq/L. Fluids will be switched to contain dextrose if the serum glucose is less than 250 mg/dL.

SUMMARY:
The purpose of this study is to determine whether adult DKA patients who present to the emergency department treated with early subcutaneous long acting insulin versus standard care receive a shorter total duration of intravenous (IV) insulin infusion.

DETAILED DESCRIPTION:
Specific Aims: To evaluate the impact of early administration of subcutaneous glargine versus standard care on time of insulin infusion in DKA patients and other secondary outcomes listed in this application.

Methods: DKA patients enrolled in this study will receive the long acting glargine dose (0.3 units/kg with a maximum dose of 30 units) within two hours after initiation the IV insulin infusion. Besides timing of the glargine dose, no other changes in standard patient care will occur in those patients enrolled in this study, the same labs will be collected and the insulin infusion will be titrated using the same hospital protocol algorithm.

Patients enrolled in the prospective arm will be compared with the retrospective control group, which received standard insulin therapy (subcutaneous insulin glargine administered at least 2 to 3 hours prior to termination of the insulin infusion). There will be 18 patients in this group selected in reverse chronological order from our pre-specified date range of 8/1/2014 to 7/31/2016.

ELIGIBILITY:
Inclusion Criteria:

* Bicarbonate <18 mg/dL
* Anion gap >16
* Blood glucose >250 mg/dL
* Ketonemia or ketonuria

Exclusion Criteria:

* Pregnant women
* Refused consent
* Patient left ED against medical advice

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Duration of intravenous insulin infusion | up to 10 months
  Measured in minutes from starting insulin infusion

SECONDARY OUTCOMES:
Time to resolution of high serum glucose (hyperglycemia) | up to 10 months
  Measured in minutes from starting insulin infusion
Time to closure of anion gap | up to 10 months
  Measured in minutes from starting insulin infusion
Time to correction of bicarbonate | up to 10 months
  Measured by serum bicarbonate
Time to correction of serum pH | up to 10 months
  Measured by pH on venous blood gas
Total duration of hospital stay | up to 10 months
  Measured in days
Return of DKA within 24 hours | up to 10 months
  Indicated by presence of diagnostic criteria within 24 hours of starting insulin infusion
Incidence of low serum glucose (hypoglycemia) within 24 hours | up to 10 months
  Measure by serum glucose.

CONTACTS AND LOCATIONS:
Overall Officials: George C Willis, MD, Principal Investigator — Director of Undergraduate Medical Education
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual subject results will not be shared with those involved in the prospective arm.